CLINICAL TRIAL: NCT02186522
Title: Immune Failure in Critical Therapy(INFECT) Study: Phenotyping Immune Cell Dysfunction to Predict Outcomes in Critically Ill Adults
Brief Title: Immune Failure in Critical Therapy (INFECT) Study
Acronym: INFECT
Status: Completed | Type: Observational
Sponsor: University of Edinburgh (Other)
Collaborators: Technology Strategy Board, United Kingdom (Other); Becton, Dickinson and Company (Industry)
Responsible Party: Sponsor
Other Study IDs: 2014/0208
Record Dates: First submitted 2014-07-07; First posted 2014-07-10 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2015-11

CONDITIONS: Sepsis; Septic Shock
Keywords: Sepsis; Septic shock; Critical care; Immune dysfunction; Inflammatory markers; Neutrophil; Monocyte; Tregs
MeSH Terms: conditions — Sepsis; Shock, Septic; Immune System Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Samples of serum and plasma stored frozen
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Critical Care Patients: Patients staying in the ICU for at least 48 hours, requiring external support of one or more organs (invasive ventilation, inotropes/vasopressors or renal replacement therapy) and who are not expected to die within 48 hours of study entry.

SUMMARY:
Patients admitted to intensive care units (ICU) are at high risk of developing secondary infections, and this is in part due to dysfunction or failure of their 'germ killing' functions (the immune system). Our group has recently identified three signatures of immune system failure which can be readily detected on a blood sample, and importantly, appear to predict the chances of developing secondary infection. Such a test would have major benefits for the management of patients in intensive care if it can be translated into a test usable in everyday clinical practice. This study aims to validate our original findings in a cohort of patients from multiple ICUs, using a test which will be suitable for everyday clinical practice, and thus take the next step towards developing a market-ready test.

Study hypothesis:

Measurement of neutrophil CD88, monocyte HLA-DR and percentage Tregs will accurately predict the risk of nosocomial infection.

ELIGIBILITY:
Inclusion Criteria:

* Age >16 (>18 in England)
* Requiring level 3 care (i.e. requiring invasive support of respiratory system alone, or two or more other organ systems (haemofiltration, inotropes/vasopressors)
* Predicted to remain in ICU for at least 48 hours,

Exclusion Criteria:

* Not expected to survive for a further 24 hours
* Known or suspected ICU-acquired infection at time of screening (non-ICU acquired nosocomial infection - i.e. non-ICU healthcare associated infection is NOT and exclusion)
* Known inborn errors of immune function
* Immunosuppression (corticosteroids up to 400mg hydrocortisone equivalent daily dose permitted)
* HIV infection
* Pregnancy
* Previously enrolled in the study

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Critical Care patients who are expected to remain in ICU for at least 48 hours, and require the external support of one or more organs (invasive ventilation, inotropes/vasopressors or renal replacement therapy) and who are not expected to die within 48 hours of study entry.
Sampling Method: Probability Sample
Enrollment: 168 (Actual)
Dates: Start 2014-07; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
The development of immune dysfunction (see below) and its association with ICU-acquired infection within the 16 day study period. | Within the first 16 days

SECONDARY OUTCOMES:
ICU Outcome (lived/died) | Within first 16 days
Death from sepsis | Within first 16 days
Organ dysfunction as determined by SOFA score | Within first 14 days
Length of ICU stay | Up to 3 months (for current hospital admission only)
Duration of organ support in ICU | Within first 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Conway Morris, MD, Principal Investigator — University of Cambridge; Tim S Walsh, MD, Principal Investigator — NHS Lothian/University of Edinburgh; John Simpson, MD, Principal Investigator — Newcastle University; Alistair Roy, MD, Principal Investigator — City Hospitals Sunderland NHS Foundation Trust; Alun Brown, Principal Investigator — Guy's and St Thomas' NHS Foundation Trust; Manu Shankar-Hari, MD, Principal Investigator — Guy's and St Thomas' NHS Foundation Trust; Anthony Bateman, MD, Principal Investigator — NHS Lothian (Western General Hospital)
Locations (4):
- United Kingdom (4):
  - Royal Infirmary of Edinburgh, Edinburgh
  - Western General Hospital, Edinburgh
  - St Thomas' Hospital, London
  - Sunderland Royal Hospital, Sunderland

REFERENCES:
- [Derived] Conway Morris A, Datta D, Shankar-Hari M, Stephen J, Weir CJ, Rennie J, Antonelli J, Bateman A, Warner N, Judge K, Keenan J, Wang A, Burpee T, Brown KA, Lewis SM, Mare T, Roy AI, Hulme G, Dimmick I, Rossi AG, Simpson AJ, Walsh TS. Cell-surface signatures of immune dysfunction risk-stratify critically ill patients: INFECT study. Intensive Care Med. 2018 May;44(5):627-635. doi: 10.1007/s00134-018-5247-0. Epub 2018 Jun 7. PMID 29915941
- [Derived] Conway Morris A, Datta D, Shankar-Hari M, Weir CJ, Rennie J, Antonelli J, Rossi AG, Warner N, Keenan J, Wang A, Brown KA, Lewis S, Mare T, Simpson AJ, Hulme G, Dimmick I, Walsh TS. Predictive value of cell-surface markers in infections in critically ill patients: protocol for an observational study (ImmuNe FailurE in Critical Therapy (INFECT) Study). BMJ Open. 2016 Jul 18;6(7):e011326. doi: 10.1136/bmjopen-2016-011326. PMID 27431901